CLINICAL TRIAL: NCT06584162
Title: Subcutaneous Vedolizumab Drug De-escalation Using Therapeutic Drug Monitoring in Inflammatory Bowel Disease: a Randomized Controlled Pilot Study
Brief Title: Subcutaneous Interval Lengthening of Vedolizumab for Economic Research
Acronym: SILVER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Geert D'Haens, Prof. dr. G.R.A.M. D'Haens, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL80854.018.22
Record Dates: First submitted 2023-06-22; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Continuing subcutaneous vedolizumab every other week
- Intervention (Experimental): Therapeutic drug monitoring guided de-escalation
  Interventions: Drug: Vedolizumab Injection

INTERVENTIONS:
Drug: Vedolizumab Injection — Based on therapeutic drug monitoring, patients could be de-escalated based on a pharmacokinetic model:
  Dosing interval Trough Target 20 mg/L
  Adjust dosing interval to:
  2 weeks < 33 mg/L 2 weeks 2 weeks 33 - 46 mg/L 3 weeks 2 weeks ≥ 46 mg/L 4 weeks 3 weeks < 20 mg/L 2 weeks 3 weeks 20 - 29 mg/L 3 weeks 3 weeks ≥ 29 mg/L 4 weeks 4 weeks < 13 mg/L 2 weeks 4 weeks 13 - 20 mg/L 3 weeks Version number: 6.1, 24-06-2024 22 of 44 4 weeks ≥ 20 mg/L 4 week
  Arms: Intervention

SUMMARY:
Rationale: Subcutaneous vedolizumab is an effective maintenance therapy for patients with inflammatory bowel disease. Patients using subcutaneous vedolizumab (every 2 weeks) have higher vedolizumab serum trough concentrations than those who are treated with intravenous vedolizumab (every 4-8 weeks). Since biologic therapies such as vedolizumab are expensive, lengthening of the injection interval (de-escalation) is of interest to reduce health care costs. However, maintaining remission while extending vedolizumab injection intervals has not been evaluated yet but represents a critical component of both medical and societal costs. Studies have suggested that higher vedolizumab serum concentrations are associated with superior clinical outcomes. Our strategy is to administer subcutaneous vedolizumab with prolonged intervals using therapeutic drug monitoring, i.e. dose based on vedolizumab concentrations, to reduce medical and societal costs while preserving remission.

Objectives: To evaluate whether subcutaneous vedolizumab therapeutic drug monitoring (TDM)-guided de-escalation will be cost-effective, compared to normal dosing regimen in patients with inflammatory bowel disease in remission. The secondary objective is to investigate the efficacy of TDM-guided de-escalation subcutaneous vedolizumab dosing compared to standard dosing.

Study design: This is a single-centre, randomized controlled, open-label pilot study.

Study population: 40 patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis) in steroid-free clinical and biochemical remission with subcutaneous vedolizumab maintenance therapy of 108 mg every other week for at least 6 months.

Intervention: Patients will be randomized (1:1) to the 'TDM-guided subcutaneous vedolizumab de-escalation' strategy versus 'standard care' (e.g. continuing standard subcutaneous vedolizumab dosing regimen of 108 mg every other week).

Main study parameters/endpoints: Primary endpoint: cost-effectiveness of the TDM-guided de-escalation group compared to the standard dosing group over 48 weeks. Secondary endpoints include: proportion of patients with sustained clinical remission (based on Harvey-Bradshaw Index or Simple Clinical Colitis Activity Index), proportion of patients with (sustained) biochemical remission (based on c-reactive protein and fecal calprotectin), pharmacokinetic differences (vedolizumab levels and immunogenicity), safety and quality of life (measured by SIBDQ and EQ-5D-5L).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease or ulcerative colitis
* Clinical and biochemical remission: absence of active inflammatory intestinal symptoms, fecal calprotectin <250 ug/g and CRP <5 mg/g, HBI <5 or SCCAI <4
* Steroid free remission for at least 6 months whilst being treated with subcutaneous vedolizumab at a stable dose of 108mg every other week.

Exclusion Criteria:

* Absence of written informed consent;
* Presence of anti-drug antibodies against vedolizumab, these levels will be determined in case the vedolizumab concentration is below 1 ug/ml;
* Concomitant oral glucocorticosteroid usage;
* Imminent need for IBD-related surgery as judged by the treating clinician;
* Actively draining peri-anal fistula;
* Patients with short bowel syndrome, an ostomy or a symptomatic stricture;
* Active participation in another interventional trial;
* Pregnancy or lactation;
* Other significant medical conditions that might interfere with this study (such as current/recent malignancy, immunodeficiency syndromes and psychiatric illness);
* Impossibility to measure outcomes, e.g. planned relocation, language issues, short life expectancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Cost-effectiveness | 48 weeks
  Medical and societal expenses will be measured troughout the study. The primary outcome is at the end of the study at Week 48. Cost-effectiveness will be measured by using a cost-questionnaire developed with the health economics department, including health-related, work-related and societal costs.

SECONDARY OUTCOMES:
Difference in Quality of Life | multipe times between baseline and 48 weeks
  Quality of life will be measured by EQ-5D-5L questionnaire
Biochemical parameters | multipe times between baseline and 48 weeks
  CRP
Biochemical parameters | multipe times between baseline and 48 weeks
  Fecal calprotectin
Pharmacokinetic aspects | multipe times between baseline and 48 weeks
  Vedolizumab concentrations
Pharmacokinetic aspects | multipe times between baseline and 48 weeks
  Anti-drug antibodies
Difference in Quality of Life | multipe times between baseline and 48 weeks
  Quality of life will be measured by SIBDQ
Clinical outcomes | multipe times between baseline and 48 weeks
  Clinical outcomes will be measured troughout the study. For ulcerative colitis patients: Simple Clinical Colitis Activity Index.
Clinical outcomes | multipe times between baseline and 48 weeks
  Clinical outcomes will be measured troughout the study. For Crohn's disease patients: Harvey-Bradshaw Index.

CONTACTS AND LOCATIONS:
Overall Officials: G.R.A.M. D'Haens, MD PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No